CLINICAL TRIAL: NCT03578835
Title: Bloodstream Infection Due to Multidrug-Resistant Organisms - Multicenter Study on Determinants of Clinical Outcomes
Acronym: BLOOMY-COM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Freiburg (Other); University Hospital Lübeck (Other); University Hospital of Berlin (Other); University of Giessen (Other); Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Prof. Dr. Evelina Tacconelli, Prof. Infectious Diseases, FESCMID,ESCMID Education Officer,EUCIC Chair, University Hospital Tuebingen
Other Study IDs: DZIF TTU 08.810
Record Dates: First submitted 2018-04-11; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Bloodstream Infection; Septic Shock
Keywords: BSI; SF-36; Clinical Outcome; Whole Genome Sequencing; Predictive Score; Bloodstream Infection; Septic Shock; Multi-resistant Bacteria
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Bacterial strains isolated from blood cultures and samples derived thereof (such as purified DNA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multi-center BSI cohort: Patients from six German study centers suffering from bloodstream infection caused by specific target organisms.

SUMMARY:
Continual surveillance of both community-acquired and nosocomial bloodstream infections for specific target organisms. Analysis of comorbidities, complications, bacterial resistance patterns, bacterial genomics (e. g. via WGS and MLST typing) for the determinants of clinical outcomes. The clinical outcomes are investigated both in the short-term (up until discharge) and the long-term (six months after index blood culture by standardized questionnaire). A predictive point-of-care score is to be developed based on these data to define high-risk patient populations requiring more intensive diagnostic and/or treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Informed consent given either by patient or guardian
* Inpatient
* At least one blood culture positive for one of the following bacteria: Staphylococcus aureus, Enterococcus spp., Escherichia coli, Enterobacter spp., Klebsiella spp., Acinetobacter baumannii, Pseudomonas aeruginosa

Exclusion Criteria:

* Less than 18 years old
* Not capable of giving informed consent nor informed consent given by guardian
* Outpatient
* No blood cultures positive for any of the target organisms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients with at least one blood culture positive for any of the target organisms: Staphylococcus aureus, Enterococcus spp., Escherichia coli, Enterobacter spp., Klebsiella spp., Acinetobacter baumannii, Pseudomonas aeruginosa.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Short-term mortality due to bloodstream infection | From index blood culture to discharge, an average of 16 days
  Mortality due to bloodstream infection up to hospital discharge in association to causative species, resistance pattern, comorbidities, complications etc.
Long-term mortality due to bloodstream infection | Up to 6 months
  Mortality due to bloodstream infection up to long-term follow-up after 6 months in association to causative species, resistance pattern, comorbidities, complications etc.
Long-term morbidity due to bloodstream infection | At 6 months
  Morbidity as measured by the SF-36 questionnaire due to bloodstream infection after 6 months in association to causative species, resistance pattern, comorbidities, complications etc.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Universitätsklinikum Tübingen, Tübingen, Bade-Württemberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Justus-Liebig-Universität Gießen, Giessen, Hesse
  - Universitätskliniken Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin, Berlin